CLINICAL TRIAL: NCT04702412
Title: Implementation of an Electronic Patient-reported Measure of Barriers to Antiretroviral Therapy Adherence With the Opal Patient Portal: a Mixed Method Type 3 Hybrid Pilot Study at a Large Montreal HIV Clinic
Brief Title: Electronic Capture of Adherence Barriers for HIV Care
Acronym: CTNPT039
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: CIHR Canadian HIV Trials Network (Network)
Responsible Party: Principal Investigator, Dr. Bertrand Lebouche, Clinical Scientist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2021-7190
Record Dates: First submitted 2020-12-11; First posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: HIV Infections
Keywords: patient-reported outcomes; adherence; antiretroviral therapy; mHealth; smartphone app; patient portal; implementation science; care
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: Pilot study with a mixed method type 3 implementation-effectiveness hybrid design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Opal patient portal (Experimental): Exposure to routine use of a patient portal (Opal) through which HIV patients are expected to complete a measure on barriers to ART adherence for screening purposes, before each HIV care visit.
  Interventions: Other: The Opal patient portal and smartphone application combined with the I-Score patient-reported outcome measure

INTERVENTIONS:
Other: The Opal patient portal and smartphone application combined with the I-Score patient-reported outcome measure — HIV patients will complete the I-Score PROM via Opal (patient portal) prior to three consecutive clinic visits with their HIV physician who is expected to access their PROM results in time for the visit. The clinic visits will be held at Time 1, Time 2 (3 months) and Time 3 (6 months).

SUMMARY:
Adherence to antiretroviral therapy (ART) remains problematic. Our team has thus developed a new patient-reported measure of barriers to ART adherence (the I-Score) which will be completed by HIV patients through the Opal patient portal for routine HIV care. This 6-month mixed method pilot study will implement the I-Score/Opal intervention with 5 HIV physicians at the McGill University Health Centre (Montreal, Quebec) and 30 of their patients. The study's primary objectives are to assess patient and physician perceptions of the intervention (e.g., acceptability) and evaluate the implementation strategy. The data collected will help plan and determine the feasibility of a definitive effectiveness trial.

DETAILED DESCRIPTION:
Background: Adherence to antiretroviral therapy (ART) remains problematic. Regular monitoring of its barriers is clinically recommended, however, patient-provider communication around adherence is often inadequate. Our team thus decided to develop a new electronically administered patient-reported outcome measure (PROM) of barriers to ART adherence (the I-Score) to facilitate the systematic capture of this data for physician consideration in routine HIV care. To prepare for a controlled definitive trial to test the I-Score intervention, a pilot study was designed. Its primary objectives are to evaluate patient and physician perceptions of the I-Score intervention and its implementation strategy.

Methods: This one-arm, 6-month study will adopt a mixed method type 3 implementation-effectiveness hybrid design and be conducted at the Chronic Viral Illness Service of the McGill University Health Centre (Montreal, Canada). Five HIV physicians and 30 of their HIV patients with known or suspected adherence problems will participate. The intervention will involve having patients complete the I-Score in the Opal smartphone application, before meeting with their physician. Both patient and physician will have access to the I-Score results, for consideration during the clinic visits at Times 1, 2 (3 months), and 3 (6 months). The implementation strategy will focus on stakeholder involvement, education, and training; promoting the intervention's adaptability; and hiring an Application Manager to facilitate implementation. Implementation, patient, and service outcomes will be collected (Times 1-2-3). The primary outcome is the intervention's acceptability to patients and physicians. Qualitative data obtained, in part, through physician focus groups (Times 2-3) and patient interviews (Times 2-3) will help evaluate the implementation strategy and inform any methodological adaptations.

Discussion: This study will help plan a definitive trial to test the efficacy of the I-Score intervention. It will generate needed data on electronic PROM interventions in routine HIV care that will help improve understanding of conditions for their successful implementation.

ELIGIBILITY:
Inclusion Criteria:

* be aged 18 years or older
* be diagnosed with HIV-1 infection
* be treated with a combination antiretroviral therapy (composed of 2 to 3 different drugs)
* be treated for HIV at the Chronic Viral Illness Service of the McGill University Health Centre
* be able to speak and understand either French or English
* possess a smartphone
* be willing to download the smartphone app

Exclusion Criteria:

* are participating in a clinical trial at the time of enrollment in this study
* have a cognitive impairment or medical instability that prevents them from participating in the interview
* have insufficient mastery of French or English to participate in the interview and complete the questionnaires
* have insufficient ability to use the app with the technical support provided
* are co-infected with hepatitis C and are being treated for it or have completed treatment 3 months or less ago
* are co-infected with hepatitis B and are either not treated for it or are being treated for it with a medication other than their anti-HIV medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the Intervention as assessed with the Acceptability E-scale | Change from baseline (week 1) to study completion (week 24)
  Score range: 6-30 (Threshold: M ≥ 24, indicates high acceptability)
Acceptability of the Intervention as indicated by the percent likely to recommend the I-Score | Change from baseline (week 1) to study completion (week 24)
  (Threshold: ≥ 80 percent)
Acceptability of the Intervention as assessed with the Net Promoter Score | Change from baseline (week 1) to study completion (week 24)
  Score range: -100 to 100 (Threshold: > 0, indicates acceptability)

SECONDARY OUTCOMES:
Appropriateness of the Intervention as assessed with the Perceived Compatibility subscale | Change from baseline (week 1) to study completion (week 24)
  Score range: 1 to 7 (Threshold: Score M ≥ 5.5, indicates high compatibility)
Appropriateness of the Intervention as assessed with the Appropriateness of Intervention Measure | Change from baseline (week 1) to study completion (week 24)
  Score range: 1 to 5 (Threshold: Score M ≥ 4, indicates high appropriateness)
Feasibility of the Intervention as indicated by the consent rate | At baseline
  Reasons for refusal will also be collected (Threshold: ≥ 70 percent)
Feasibility of the Intervention as indicated by the retention rate | Cumulative until study completion (week 24)
  (Threshold: ≥ 80 percent)
Feasibility of the Intervention as indicated by the missing I-Score data rate | Cumulative until study completion (week 24)
  e.g., due to non-completion, network failure (Threshold: ≤ 10 percent)
Feasibility of the Intervention as assessed with the Feasibility of Intervention Measure | Change from baseline (week 1) to study completion (week 24)
  Score range: 1 to 5 (Threshold: M ≥ 4, indicates high feasibility)
Fidelity of the Intervention as indicated by the percentage of patients who complete the I-Score on time | Cumulative until study completion (week 24)
  (Threshold: ≥ 90 percent)
Fidelity of the Intervention as indicated by the percentage of physicians who review the I-Score results on time | Cumulative until study completion (week 24)
  (Threshold: ≥ 90 percent)
Feasibility of the implementation strategy as indicated by the percentage of physicians who participate in the implementation activities | Cumulative until study completion (week 24)
  e.g., educational meeting, focus groups (Threshold: ≥ 80 percent)
Feasibility of the implementation strategy as indicated by the number of technical issues encountered | Cumulative until study completion (week 24)
  Based on the Application Manager's notes

OTHER OUTCOMES:
Patient management as indicated by the proportion of clinical visits where physicians took action based on I-Score results | Change from baseline (week 1) to study completion (week 24)
  Only among visits that identified an adherence barrier of concern with the I-Score PROM
Barriers to ART adherence as measured by the I-Score PROM | Change from baseline (week 1) to study completion (week 24)
  Score range: 1 to 20, where higher scores indicate a greater number of problematic barriers
Adherence to ART as measured by the Self-Rating Scale Item | Change from baseline (week 1) to study completion (week 24)
  Score range: 1 to 6, where higher scores indicate higher adherence
HIV RNA viral load as indicated in the patient's medical file | Change betweem baseline (week 1) and study completion (week 24)
  Range: Detectable, where > 50 copies/mL = detectable, an undesirable clinical outcome, or Undetectable

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Lebouché, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Research Institute of the McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Engler K, Ahmed S, Lessard D, Vicente S, Lebouche B. Assessing the Content Validity of a New Patient-Reported Measure of Barriers to Antiretroviral Therapy Adherence for Electronic Administration in Routine HIV Care: Proposal for a Web-Based Delphi Study. JMIR Res Protoc. 2019 Aug 2;8(8):e12836. doi: 10.2196/12836. PMID 31376275
- [Background] Lessard D, Engler K, Toupin I; I-Score Consulting Team; Routy JP, Lebouche B. Evaluation of a project to engage patients in the development of a patient-reported measure for HIV care (the I-Score Study). Health Expect. 2019 Apr;22(2):209-225. doi: 10.1111/hex.12845. Epub 2018 Oct 29. PMID 30375111
- [Background] Kildea J, Battista J, Cabral B, Hendren L, Herrera D, Hijal T, Joseph A. Design and Development of a Person-Centered Patient Portal Using Participatory Stakeholder Co-Design. J Med Internet Res. 2019 Feb 11;21(2):e11371. doi: 10.2196/11371. PMID 30741643
- [Derived] Engler K, Vicente S, Ma Y, Hijal T, Cox J, Ahmed S, Klein M, Achiche S, Pant Pai N, de Pokomandy A, Lacombe K, Lebouche B. Implementation of an electronic patient-reported measure of barriers to antiretroviral therapy adherence with the Opal patient portal: Protocol for a mixed method type 3 hybrid pilot study at a large Montreal HIV clinic. PLoS One. 2021 Dec 30;16(12):e0261006. doi: 10.1371/journal.pone.0261006. eCollection 2021. PMID 34969046